CLINICAL TRIAL: NCT06130605
Title: Subjects Perceived as Embarrassing During a Consultation in General Medical Practice
Acronym: Gene-MG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_006_Gene-MG
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: General Practice
Keywords: general medical consultation; gene; modesty; fear of judgment
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- people over the age of 18: people over the age of 18.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Optimal medical care requires transparency and honesty. However, it is not always easy to address some issues that may be considered too personal, intimate or taboo, such as mental health, sexuality, addiction and death. Patients' approach to these issues may be influenced by the profile of their general practitioner, or by the atmosphere of the consultation.

This retention of information by the patient, whether voluntary or not, can lead to adverse events related to care due to a misunderstanding between doctor and patient.

DETAILED DESCRIPTION:
The main objective is to describe the proportion of patients limiting the subjects addressed during a general medicine consultation by gene, modesty and/or fear of judgment The secondary objective is to study the factors associated with limitation of subjects addressed by patient by gene, modesty and/or fear of judgment during a general medicine consultation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Agreeing to take part in the study

Exclusion Criteria:

* Minors
* Protected by law (guardianship, curatorship, safeguard of justice)
* Refusing to take part in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people over the age of 18 agreeing to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
limitation of subjects addressed by gene, modesty and/or fear of judgment | Day 0
  Proportion of patients who have ever restricted the subjects discussed during a general medical consultation by gene, modesty and/or fear of judgment

CONTACTS AND LOCATIONS:
Overall Officials: THERY MERLAND Emilie, Dr, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided